CLINICAL TRIAL: NCT00427063
Title: Heredity of Retinal Vessel Tortuosity - A Twin Study
Brief Title: Heredity of Retinal Vessel Tortuosity
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Other Study IDs: Danish Twin Registry 1998
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Retinopathy of Prematurity
Keywords: retinal vessels; tortuosity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to asses the relative influence of genetic and environmental influence on the tortuosity of retinal arterioles in eyes of 218 healthy Danish twins aged 20-46 years. We expect to find a high heredity for the variation in tortuosity. This knowledge can contribute to the elucidation of the pathology in retinal diseases.

DETAILED DESCRIPTION:
All persons underwent an ophthalmic examination including refraction, slit lamp biomicroscopy and digital fundus photography. Two independent graders (both with an MD degree) made a visual grading of the severity of tortuosity of the retinal arterioles in the fundus images.

ELIGIBILITY:
Inclusion Criteria:

* Samesex twin pairs of self-assessed good health

Exclusion Criteria:

* Diabetes mellitus
* Hypertension
* Thyroid disease
* Cataract or other opacities of the refractive media
* Missing fundus photographs

Ages: 20 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218
Dates: Start 1998-01; Study Completion 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larsen, Prof. MD, Principal Investigator — Department of Ophthalmology Glostrup Hospital University of Copenhagen
Locations (1):
- Department of Ophthalmology Glostrup Hospital, Glostrup Municipality, Copenhagen County, Denmark